CLINICAL TRIAL: NCT04926857
Title: DEFINE AFib Atrial Fibrillation - Development of a Predictive Model for Future Health Care Utilization From Measurements Collected From an Implantable Cardiac Monitor.
Brief Title: DEFINE AFib (Atrial Fibrillation)
Acronym: DEFINE AFib
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20024
Record Dates: First submitted 2021-01-04; First posted 2021-06-15 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
DEFINE AFib is a prospective, observational, post-market clinical study administered to patients via the Medtronic Discovery app platform. This study will enroll approximately 5,000 patients in the United States who have a Reveal LINQ or LINQ II ICM (or future market-released LINQ devices) and an Apple® iPhone® with iOS version 13 or higher. Interested participants will be screened through the Medtronic Discovery app and those eligible will complete an app-based informed consent. Participants will receive health-focused and quality of life surveys at variable timepoints. DEFINE AFib will measure healthcare interactions using administered surveys to identify said interactions. The Medtronic Discovery app will provide participants with a summary of their ICM data. Participants will be followed up to 5 years or to the end of their ICM service life.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the association between complex patterns of device-detected AF and other summary and episodic measurements collected by the market- released LINQ ICM device and AF-related healthcare utilization, quality of life, AF-related symptoms, and specific clinical outcomes in patients with a market-released LINQ ICM. The Medtronic Discovery app will be used to collect data both (1) via the iPhone® through patient-reported health surveys and Bluetooth-enabled devices connected through the Apple Health app and (2) data accessed through or stored on the phone pertaining to health records, activity, and other lifestyle data. Secondarily, this study will examine associations between clinical procedures, medications and lifestyle actions taken and their impact on device-detected AF. Additionally, this study will help Medtronic evaluate patients' interaction with reports generated from health data collected by the market-released LINQ ICM. This study will improve our understanding of how data from the LINQ family of devices can be used to guide the management of AF patients.

ELIGIBILITY:
Inclusion Criteria

* Patients with a LINQ ICM who have a self-reported history of AF and who have received an ICM for the following device-logged indications, categorized into the following discrete groups:

  * AF management: AF management and post-ablation management indications
  * Suspected AF: Suspected AF and palpitations indications
  * Stroke: Cryptogenic stroke indication
* Individual Access and ability to use an Apple iPhone® compatible with Medtronic's research app (iOS® v. 13.X or higher)
* Patient is willing and able to comply with the protocol, including CareLink transmissions (requires adequate connectivity), remotely administered instructions, and remote survey participation
* Patient is 22 years of age or older
* Located in the United States, with CareLink managed through servers located in United States (50 states or District of Columbia)
* Valid email address from self-report at enrollment
* Patient must be able to read and write in English

Exclusion Criteria Patients with > 24 months elapsed time from recorded LINQ device implant or > 48 months elapsed from recorded LINQ II implant date

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Atrial Fibrillation and a LINQ device
Sampling Method: Non-Probability Sample
Enrollment: 973 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Piccini, MD, Principal Investigator — Duke University
Locations (26):
- United States (26):
  - Saint Joseph Heritage Hospital, Mission Viejo, California
  - Desert Heart Rhythm Consultants, Palm Springs, California
  - Florida Electrophysiology Associates, Atlantis, Florida
  - Cardiac Arrhythmia Service, Boca Raton, Florida
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - HCA Healthcare, Overland Park, Kansas
  - Stormont Vail Health Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Norton Heart Specialists, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Huntington Hospital, Huntington, New York
  - NYU Langone Hospital Long Island, Mineola, New York
  - White Plains Hospital Medical Center, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health, Greensboro, North Carolina
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - St. Luke's Cardiology Associates, Bethlehem, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Ascension Seton Heart Institute Clinical Research, Austin, Texas
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During study execution, there was a sponsor decision to end the study earlier, so the study enrolled far less than the 5000 enrollments specified by the protocol.
Groups:
- Enrolled Patients: Patients that completed a survey on the study App that confirmed that they met the inclusion/exclusion criteria of the study and that they read and agreed with the informed consent.
Period: Overall Study
Arm/Group | Enrolled Patients
Started | 973
Completed | 864
Not Completed | 109
Not completed — Withdrawal by Subject | 40
Not completed — Death | 9
Not completed — Study product no longer in use | 44
Not completed — Inadequate data to address primary objective | 16

BASELINE CHARACTERISTICS:
Population: Due to eligibility survey responses permanently missing for 3 subjects, 970 of the 973 subject enrollments are included in all analysis.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 970
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 276
  >=65 years | 694
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 414
  Male | 556
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 777
  More than one race | 22
  Unknown or Not Reported | 136
Region of Enrollment [Number; unit: participants]
  United States | 970
Reason for enrollment [Count of Participants; unit: Participants] — Patients in the study received a LINQ device for one of the following reasons: AF ablation, AF management, cryptogenic stroke, palpitations or suspected AF
  Participants
    AF Management | 584
    AF Ablation | 181
    Cryptogenic Stroke | 91
    Palpitations | 20
    Suspected AF | 94

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Utilization Where AF Was a Reason or a Suspected Reason for the Healthcare Interaction.
Description: Primary objective is to evaluate whether summary and episodic measurements collected by market-released LINQ ICMs are able to predict increased AF-related healthcare utilization (HCU), which are confirmed healthcare visits in the inpatient hospital, outpatient hospital, clinic/office, emergency department, or other care location (including remote visits) where AF was a reason or suspected reason for healthcare interaction.
  A predictive model was trained on 70% of the patients with adequate data available and assessed in a validation data set of the remaining 30% of patients, using rolling 60 day blocks. In each block, measurements in the first 30 days were used to predict whether confirmed HCU occurred in the trailing 30 days. Predictive value was assessed using sensitivity, specificity and other measurements within a confusion matrix as well as an area under the receiver operator curve, balancing the sensitivity and specificity. Outcome measure entered here will be AUROC.
Time Frame: Through study completion (2 years of enrollment, up to 2.6 years of follow-up)
Measure: Number (95% Confidence Interval); unit: Proportion
Groups:
- Training and Testing Partitions: The set of enrolled patients that had enough device follow-up for a lead-in portion and a prediction portion was used to develop a prediction model for increase healthcare utilizations. There were 864 total patients with sufficient device follow-up. Patients were partitioned into a training set (N=601) and a testing set (N=263). A predictive model was built with the training set and assessed for predictive value in the testing set.
Arm/Group | Training and Testing Partitions
Number analyzed (Participants) | 864
Proportion | 0.76 [0.70 to 0.81]

ADVERSE EVENTS:
Time Frame: All cause mortality was monitored from time of enrollment to completion of study (up to 2.6 years of follow-up). Adverse events were not required and were not collected to meet the objectives of this study.
Description: All cause mortality was monitored, but adverse events were not required and were not collected to meet the objectives of this study.
Arm/Group | Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 9/970
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT04926857/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04926857/SAP_001.pdf